CLINICAL TRIAL: NCT05718440
Title: Individualisation of Uronephrological Complications Risk Factors in Spinal Dysraphism
Brief Title: Uronephrological Complications Risk Factors in Spinal Dysraphism
Acronym: RUD
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221008
Record Dates: First submitted 2023-01-12; First posted 2023-02-08 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Spinal Dysraphism
Keywords: spinal dysraphism; uronephrological complications; risk factors; urinary dysfunction; bowel dysfunction; sexual dysfunction
MeSH Terms: conditions — Spinal Dysraphism; Intestinal Diseases; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with spinal dysraphism
  Interventions: Other: Individualisation of uronephrological complications risk factors

INTERVENTIONS:
Other: Individualisation of uronephrological complications risk factors — description of pelvic disorders in terms of clinical presentation, electrophysiology/urodynamics/anorectal manometry patterns, urethrocystography/urinary ultrasound/defecography results and urinary complications (infections, vesicoureteral reflux), depending on the dysraphim's type and level of injury and to correlate these parameters to the uronephrological risk factors and complications recorded.

SUMMARY:
Spinal dysraphism consist of congenital malformations resulting of abnormalities in the formation of neural tube and/or surrounding structures during embryogenesis. The aim of this study is to assess if there are specific clinical and paraclinical patterns of pelvic (urinary, bowel, sexual) disorders depending on the dysraphism's type and level of injury.

This description will help to determine a prognosis on symptoms and the risk of complication depending on the dysraphism's type and level of injury. It will provide targeted evaluation and cares: identifying patients who will be at risk of complications and needing acute monitoring or preventing cares on the symptoms' onset.

Pelvic disorders have an important impact on morbi-mortality (urinary dysfunction is the first cause of mortality in adults by renal failure or infection) and also on patients' quality of life.

DETAILED DESCRIPTION:
Spinal dysraphism consist of congenital malformations resulting of abnormalities in the formation of neural tube and/or surrounding structures during embryogenesis. The aim of this study is to assess if there are specific clinical and paraclinical patterns of pelvic (urinary, bowel, sexual) disorders depending on the dysraphism's type and level of injury.

This description will help to determine a prognosis on symptoms and the risk of complication depending on the dysraphism's type and level of injury. It will provide targeted evaluation and cares: identifying patients who will be at risk of complications and needing acute monitoring or preventing cares on the symptoms' onset.

Pelvic disorders have an important impact on morbi-mortality (urinary dysfunction is the first cause of mortality in adults by renal failure or infection) and also on patients' quality of life.

This is an observational descriptive study with prospective inclusions of patients over 18 years old with spinal dysraphism, evaluated for urinary, anorectal, sexual dysfunctions in a one-day hospitalization.

Inclusions will be recorded during this one-day hospitalization. On this day, patients will have a medical consultation and data concerning medical history, treatments, pelvic disorders' characteristics and physical examination will be recorded. They will answer questionnaires on pelvic dysfunctions, quality of life, anxiety and depression, cognitive disorders and self-catheterizations' adherence or difficulties. They will also undergo urodynamics. In case of peripheral neurological pattern, a perineal electrophysiology will be done with recording of bulbocavernosus reflex latency and somatosensory evoked potentials.

Outpatient examinations (urinary ultrasound, urethrocystography, anorectal manometry, defecography blood test with serum creatinine, glycemia, TSH, lipids) will be collected at the next consultation.

Patients' participation will last 12 months maximum (time period between the one-day hospitalization (inclusion) and the follow up consultation where the outpatients' examinations results will be recorded).

A better understanding of pelvic dysfunctions, according to neurological systematization and type of spinal dysraphism, will help to focus the evaluation and therapeutic managements on patients with spinal dysraphism at risk of uronephrological complications.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 18 years old with spinal dysraphism,
* urinary and/or bowel and/or sexual dysfunction,
* evaluated in a one day consultation in a neuro-urology department.
* Informed consent is required from the patient or his tutor/curator if he is under legal protection

Exclusion Criteria:

* language barrier with non-understanding of French language,
* other neurologic pathologies except syringomyelia, Chiari malformation or hydrocephalus who are often associated to spinal dysraphism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over 18 years old with spinal dysraphism
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
sexual dysfunctions in term of spinal dysraphisms | 1 day
  Sexual dysfonctions according the scale Men Health Sexual Questionnaire (MHSQ) score between 5 to 125 (no problem)
patient quality of life | 1 day
  questionnaire "Qualiveen" (quality of life linked to health) to be completed by patient (score between 0 (no problem) to 4)
Urinary disorders | 1 day
  Urinary Symptom Profile (USP) questionnaire (score between 0 (no problem) to 39)
cognitive disorders | 1 day
  Montreal Cognitive Assessment (MOCA) scale (score between 0 to 30, normal between >=26)
pelvic disorders description thanks to exams | 1 day
  urinary echography, anorectal manometry and defecography will be performed in order to described pelvic disorders n.

SECONDARY OUTCOMES:
urinary complications | 1 day
  number of infections, vesicoureteral reflux

CONTACTS AND LOCATIONS:
Locations (1):
- Tenon hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No